CLINICAL TRIAL: NCT01919814
Title: A Short-Term Appetite Suppression Trial Using Appethyl™: The Pizza
Acronym: Pizza
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Greenleaf Medical (Unknown)
Responsible Party: Principal Investigator, Frank Greenway, Clinical Medical Doctor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: PBRC 13022
Record Dates: First submitted 2013-08-02; First posted 2013-08-09 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Appethyl™, then Placebo (Active Comparator): Participants receive Appethyl™ liquid once four hours after breakfast. After a washout period of at least one week, they received the placebo drink once four hours after breakfast.
  Interventions: Dietary Supplement: Appethyl™; Other: Placebo
- Placebo, then Appethyl™ (Placebo Comparator): Participants receive the placebo drink once four hours after breakfast. After a washout period of at least one week, they received Appethyl™ liquid once four hours after breakfast.
  Interventions: Dietary Supplement: Appethyl™; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Appethyl™ — Four hours after breakfast participants will be given a small amount of liquid to drink that will contain Appethyl™. They will not know which they are getting and it will be decided randomly, like flipping a coin. Participants will be presented with a pizza in a quantity more than they could reasonably be expected to eat 5 hours after the start of their lunch meal and be asked to eat to their satisfaction over 30 minutes. Participants are not expected to eat all of the pizza.
Other: Placebo — Four hours after breakfast, participants will be given a small amount of liquid to drink that will contain a placebo (inactive liquid). Participants will not know which they are getting and it will be decided randomly, like flipping a coin. Participants will be presented with a pizza in a quantity more than they could reasonably be expected to eat 5 hours after the start of their lunch meal and be asked to eat to their satisfaction over 30 minutes. They are not expected to eat all of the pizza.

SUMMARY:
The purpose of the study is to determine whether Appethyl™, made from spinach, will reduce appetite and hunger given on the same day of testing.

DETAILED DESCRIPTION:
Four hours after breakfast a small amount of liquid to drink will be given to a participant that will contain either the Appethyl™ or placebo. Participants will be given a lunch of about 750 calories and 40% fat prepared by the Metabolic Kitchen and be asked to eat all of it. Participants will have food choice testing performed 4 hours after starting their lunch meal. This will be done in two ways. Participants will be given a list of two foods that are made of carbohydrate like bread and pretzels and be asked which is most preferred. Participants will also be given a list of foods that differ in the amounts of fat, carbohydrate and protein that they contain and will be asked to mark the ones that appeal to them.

Participants will be presented with a pizza in a quantity more than they could reasonably be expected to eat 5 hours after the start of their lunch meal and be asked to eat to their satisfaction over 30 minutes. Participants are not expected to eat all of the pizza.

ELIGIBILITY:
Inclusion Criteria:

* You are a male or female aged 18 to 65 years.
* You have a BMI (a number calculated from your height and weight) between 25-35 kg/m2, inclusive.
* Your waist circumference is over 35 inches.

Exclusion Criteria:

* You have been on a diet for weight loss in the last 2 months.
* You are being treated for blood pressure, diabetes, heart disease, rheumatoid arthritis, or blood vessel disease.
* You have a psychotic illness.
* You have other chronic diseases like an inflammatory bowel disease such as Crohn's disease or ulcerative colitis.
* You have a dysfunction of your gastrointestinal tract.
* You have food allergies.
* You have rheumatoid arthritis with inflammation.
* You have chronic constipation.
* You are taking any products to lose weight such as medication for obesity or non-prescription medications for weight loss.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Greenway, MD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Appethyl™ First, Then Placebo: Appethyl™ liquid once four hours after breakfast.
  Appethyl™: • Four hours after breakfast participants will be given a small amount of liquid to drink that will contain Appethyl™. After one week washout period, participants were given placebo drink.
  Participants will not know which they are getting and it will be decided randomly, like flipping a coin. Participants will be presented with a pizza in a quantity more than they could reasonably be expected to eat 5 hours after the start of their lunch meal and be asked to eat to their satisfaction over 30 minutes. Participants are not expected to eat all of the pizza.
- Placebo First, Then Appethyl™: Four hours after breakfast participants will be given a small amount of liquid to drink that will contain a placebo (inactive liquid). After a one week washout period, they were given Appethyl™.
  Participants will not know which they are getting and it will be decided randomly, like flipping a coin. Participants will be presented with a pizza in a quantity more than they could reasonably be expected to eat 5 hours after the start of their lunch meal and be asked to eat to their satisfaction over 30 minutes. Participants are not expected to eat all of the pizza.
Period: Overall Study
Arm/Group | Appethyl™ First, Then Placebo | Placebo First, Then Appethyl™
Started | 30 | 30
Completed | 27 | 30
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant was dropped because of adverse event
Groups:
- All Participants: Appethyl™ liquid or Placebo once four hours after breakfast.
  Appethyl™: Four hours after breakfast participants will be given a small amount of liquid to drink that will contain Appethyl™ pr Placebo.
  Participants will not know which they are getting and it will be decided randomly, like flipping a coin. Participants will be presented with a pizza in a quantity more than they could reasonably be expected to eat 5 hours after the start of their lunch meal and be asked to eat to their satisfaction over 30 minutes. Participants are not expected to eat all of the pizza.
Arm/Group | All Participants
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 30
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Difference in Pizza Consumed During Two Meals
Description: Four hours after breakfast administration of Appethyl™ or placebo(inactive liquid) is given. You will be presented with a standard lunch and then (5 hours after lunch) pizza in a quantity of more than you could reasonably be expected to eat 5 hours after the start of your lunch meal and be asked to eat to your satisfaction over 30 minutes. You are not expected to eat all of the pizza.
Time Frame: 5 hours after lunch (9 hours after administration of Appethyl from the morning)
Population: One participant dropped because of adverse event
Measure: Mean (Standard Deviation); unit: calories
Groups:
- Appethyl™: Appethyl™ liquid once four hours after breakfast.
  Appethyl™: Four hours after breakfast participants will be given a small amount of liquid to drink that will contain Appethyl™. Participants will not know which they are getting and it will be decided randomly, like flipping a coin. Participants will be presented with a pizza in a quantity more than they could reasonably be expected to eat 5 hours after the start of their lunch meal and be asked to eat to their satisfaction over 30 minutes. Participants are not expected to eat all of the pizza.
- Placebo: Four hours after breakfast participants will be given a small amount of liquid to drink that will contain a placebo (inactive liquid). Participants will not know which they are getting and it will be decided randomly, like flipping a coin. Participants will be presented with a pizza in a quantity more than they could reasonably be expected to eat 5 hours after the start of their lunch meal and be asked to eat to their satisfaction over 30 minutes. Participants are not expected to eat all of the pizza.
Arm/Group | Appethyl™ | Placebo
Number analyzed (Participants) | 59 | 59
calories | 1020.21 (554.35) | 1067.46 (551.63)
Statistical Analysis 1: Comparison: Appethyl™ vs Placebo; Test type: Superiority; p > 0.05, t-test, 2 sided — Threshold P-Value was 0.05

2. Secondary Outcome: Evaluation of Appetite
Description: The Visual Analogue scale allows you to mark a vertical line across the horizontal scale on how hungry you are or not. The Visual Analogue scale was used to evaluate hunger, fullness, longing for food, prospective intake, satisfaction, desire for salty food, desire for savory food, thirst, and desire for sweet food. The scale ranged from 0 to 100mm; the higher values indicated greater outcomes.
Time Frame: 30 minutes, 60 minutes, 120 minutes after consuming the drug or placebo
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Appethyl™ | Placebo
Number analyzed (Participants) | 59 | 59
units on a scale
  Hunger - 30 minutes | 12.14 (29.53) | 15.77 (20.40)
  Hunger - 60 minutes | 20.42 (20.53) | 22.13 (20.31)
  Hunger - 120 minutes | 30.16 (20.53) | 37.03 (20.31)
  Fullness - 30 minutes | 85.7 (21.30) | 85.29 (21.15)
  Fullness - 60 minutes | 80.00 (21.30) | 73.51 (21.02)
  Fullness - 120 minutes | 63.74 (21.30) | 59.80 (21.02)
  Longing for Food - 30 minutes | 12.59 (20.21) | 14.27 (20.11)
  Longing for Food - 60 minutes | 17.40 (20.21) | 22.39 (20.03)
  Longing for Food - 120 minutes | 27.49 (20.21) | 34.29 (20.03)
  Prospective Intake - 30 minutes | 18.11 (22.42) | 19.19 (22.33)
  Prospective Intake - 60 minutes | 21.33 (22.42) | 26.49 (22.25)
  Prospective Intake - 120 minutes | 34.48 (22.42) | 39.70 (22.25)
  Satisfaction - 30 minutes | 82.67 (23.28) | 81.76 (23.11)
  Satisfaction - 60 minutes | 72.41 (23.28) | 70.65 (22.98)
  Satisfaction - 120 minutes | 57.94 (23.28) | 53.16 (22.98)

3. Secondary Outcome: Evaluation of Satiety by Means of Visual Analogue Scale
Description: as for outcome 2
Time Frame: 30 minutes, 60 minutes, 120 minutes after consuming the drug or placebo
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Appethyl™ | Placebo
Number analyzed (Participants) | 59 | 59
units on a scale
  Desire for Salty Food - 30 minutes | 26.28 (28.20) | 30.53 (28.16)
  Desire for Salty Food - 60 minutes | 28.53 (28.20) | 34.59 (28.12)
  Desire for Salty Food - 120 minutes | 35.51 (28.20) | 40.62 (28.12)
  Desire for Savory Food - 30 minutes | 34.34 (30.75) | 38.83 (30.68)
  Desire for Savory Food - 60 minutes | 34.16 (30.75) | 40.63 (30.62)
  Desire for Savory Food - 120 minutes | 44.58 (30.75) | 46.31 (30.62)
  Thirst - 30 minutes | 27.76 (26.38) | 35.61 (26.29)
  Thirst - 60 minutes | 37.63 (26.38) | 43.01 (26.21)
  Thirst - 120 minutes | 47.69 (26.38) | 52.92 (26.21)
  Desire for Sweet Food - 30 minutes | 43.32 (32.45) | 47.75 (32.34)
  Desire for Sweet Food - 60 minutes | 47.50 (32.45) | 48.77 (32.24)
  Desire for Sweet Food - 120 minutes | 53.58 (32.45) | 53.38 (32.24)

ADVERSE EVENTS:
Arm/Group | Appethyl™ | Placebo
Serious Adverse Events (participants affected / at risk) | 1/60 | 1/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Appethyl™ (N=60) | Placebo (N=60)
Severe Headache (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No